CLINICAL TRIAL: NCT07395323
Title: Impact of Using a Virtual Reality Application on the Sleep Quality of Caregivers Working Night Shifts
Brief Title: Impact of Relaxation Sessions Using a Virtual Reality Application on the Sleep Quality of Caregivers Working Night Shifts
Acronym: Luciole
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: D24-P018
Record Dates: First submitted 2025-12-22; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-11

CONDITIONS: Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: Arm 1: Experimental (VR)
  Intervention: Virtual reality sessions
  Description: Participants undergo virtual reality sessions during this period.
  Arm 2: Control (No VR)
  Intervention: No virtual reality or standard care
  Description: Participants do not undergo virtual reality sessions during this period.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control comparator. (Active Comparator): The participant receives the actigraph again and maintains their usual bedtime and sleep-onset routine, completing the paper sleep diary for sleep quality after each waking.
  The PSQI scale is measured on the first day (D1) and again after the last night (D30).
  The sleep-wake rhythm will be analyzed using an actimeter.
  Interventions: Device: Arm 2: Control (No VR / Standard Care)
- Arm 1: Experimental (VR) (Experimental): Intervention: Virtual reality sessions
  Description: Participants undergo virtual reality sessions during this period. The sleep-wake rhythm will be analyzed using an actimeter. The sleep-wake rhythm will be analyzed using an actimeter.
  Interventions: Device: Arm 1: Experimental (VR) Intervention: Virtual reality sessions

INTERVENTIONS:
Device: Arm 1: Experimental (VR) Intervention: Virtual reality sessions — During the virtual reality period (1 month), the participant receives a VR headset and an actigrapher, provided by a Registered Nurse Practitioner (RNP). A training session is organized and scheduled following enrollment. The participant will keep the VR headset and actigrapher at home for one month. The devices will be collected by the night shift supervisor at the end of the usage period. A paper sleep diary will be provided to assess sleep quality.
  Arms: Arm 1: Experimental (VR)
Device: Arm 2: Control (No VR / Standard Care) — Intervention: No virtual reality or standard care
  Description: Participants do not undergo virtual reality sessions during this period.
  The sleep-wake rhythm will be analyzed using an actimeter.
  Arms: control comparator.

SUMMARY:
This project aims to evaluate the impact of relaxation sessions conducted using a virtual reality device on the sleep quality of night-shift healthcare workers. The intervention specifically targets the immediate post-night-shift period, a critical time for recovery, by offering immersive guided relaxation experiences designed to reduce anxiety and promote both mental and physiological relaxation.

DETAILED DESCRIPTION:
Paramedical staff working night shifts are particularly exposed to sleep disorders and psychological difficulties due to the length and organization of their working hours. The ANSES report highlights the central role of anxiety, both as a consequence of night work and as a factor that worsens sleep disturbances.

In response to this situation, the GHU Directorate of Nursing, in collaboration with Occupational Health, the CHRONOS team, and the pain specialist physician, has initiated a reflection on preventive actions aimed at better addressing the vulnerability of healthcare professionals. The objective is to provide concrete responses to psychological distress and the high levels of stress experienced by healthcare workers, which have been further intensified by the health crisis.

Within this framework, it is proposed to specifically address immediate post-night-shift sleep disturbances by implementing a relaxation program using a virtual reality application. This non-pharmacological approach aims to reduce anxiety and improve recovery among paramedical professionals working night shifts.

ELIGIBILITY:
Inclusion Criteria:

* State-certified nurse or nursing assistant (GHU, GHPG staff)
* Regularly working night shifts and on duty in the units
* Age 18 years and over
* Informed individuals who have signed written consent
* Individuals affiliated with a social security scheme and must be able to understand and read French.

Exclusion Criteria:

* No possibility of follow-up (subjects on fixed-term contracts, ongoing transfers, student reinforcements, etc.)
* Subjects with insufficient command of the French language, preventing them from taking the tests
* Pregnant or breastfeeding women (disruption of the sleep cycle), or women with young children.
* Individuals with a pacemaker or any other implanted medical device, unless medically advised otherwise (due to the radio-magnetic waves emitted by the virtual reality headset)
* Individuals with epilepsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Compare the evolution of sleep quality of paramedical professionals assessed by the PSQI scale, with or without intervention, (cross-over design). | 15 months
  The PSQI provides a score ranging from 0 to 3 for each of the seven components, as well as an overall sleep quality score ranging from 0 to 21, with higher scores indicating poorer sleep quality.
  The PSQI self-administered questionnaire is used in research and clinical practice to assess sleep quality before and after pharmacological treatment or behavioral therapy in order to measure the impact of the intervention on individuals' sleep.

SECONDARY OUTCOMES:
Severity of sleep disorders: ISI, | 15 months
  Score Total: 0 to 28
  Interpretation
  0-7: No clinically significant insomnia
  8-14: Mild insomnia (subthreshold)
  15-21: Moderate insomnia
  22-28: Severe insomnia
Level of Anxiety: GAD-7 | 15 months
  Interpretation
  0-4: Minimal anxiety
  5-9: Mild anxiety
  10-14: Moderate anxiety
Level of anxiety and depression: QIDS | 15 months
  Total: 0 to 27
  Interpretation
  0-5: No depression
  6-10: Mild depression
  11-15: Moderate depression
  16-20: Severe depression
  21-27: Very severe depression

OTHER OUTCOMES:
Work-related quality of life: PROQOL 5 | 15 months
  The scale consists of 30 items, rated on a 5-point Likert scale ranging from 1 (Never) to 5 (Very often).
  It measures three distinct dimensions (10 items each):
  Compassion Satisfaction (CS)
  - Pleasure and fulfillment derived from being able to do one's work well.
  Burnout (BO) - Feelings of exhaustion, frustration, anger, and depression related to work.
  Secondary Traumatic Stress (STS)
  - Work-related exposure to extremely stressful or traumatic events experienced by others.
  Each subscale is scored separately.
Overall quality of life: Duke Health Profile | 15 months
  The Duke Health Profile (DUKE) is a generic self-administered questionnaire designed to measure perceived health status and overall quality of life in adults. It is brief, easy to administer, and widely used in clinical and research settings.
  The questionnaire consists of 17 items, assessing health over the previous week. Responses are scored and transformed to a 0-100 scale.
Participant satisfaction: Visual Analog Scale (VAS) | 15 months
  Score: 0-100 mm
  Description:
  Participant satisfaction is assessed using a Visual Analog Scale (VAS), which consists of a horizontal line, typically 100 mm in length, anchored at each end by two extremes:
  0: Not satisfied at all
  100: Extremely satisfied
  Interpretation:
  Low scores → Low level of satisfaction
  Intermediate scores → Moderate satisfaction
Severity of sleep disorders: ESS | 15 months
  Score Total: 0 to 24
  Interpretation
  0-10: Normal
  11-15: Moderate excessive sleepiness
  ≥16: Severe excessive sleepiness
Severity of sleep disorders: NSI | 15 months
  Score Total: 0 to 20
  Interpretation: Higher scores indicate more frequent and debilitating nightmares. Often used in connection with PTSD, anxiety, and depression.
Severity of sleep disorders: MCTQ | 15 months
  Content
  Bedtime, sleep onset time, and wake-up time
  Distinction between workdays and free days
  Main score
  MSF (Mid-Sleep on Free days)
  MSFsc (Mid-Sleep on Free days, sleep-corrected)
  Interpretation
  An earlier MSFsc indicates a morning chronotype

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie results in publication could be shared. IPD detailed in the protocol of a planned metaanalysis could be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the last publication
Access Criteria: Data sharing must be accepted by the sponsor and the PI. Technical feasibility and financial support will be discussed before mandatory contractualization. Processing of shared data must comply with GDPR.